CLINICAL TRIAL: NCT05803252
Title: Videoconferencing-based Focused Acceptance and Commitment Therapy for Parents of Children With Special Health Care Needs: A Non-randomised Controlled Feasibility Trial
Brief Title: Videoconferencing-based Focused Acceptance and Commitment Therapy for Parents of SHCN Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Christian Service (Other); Hong Kong Federation of Youth Groups (Unknown); Hong Kong Young Women's Christian Association (Other); Yang Memorial Methodist Social Service (Other)
Responsible Party: Principal Investigator, Yuen Yu CHONG, Assistant Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTEC-2023-058
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Neurodevelopmental Disorders; Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder; Development Delay; Chronic Disease
Keywords: Special health care needs (SHCN); Parental well-being; Family functioning; Acceptance and Commitment Therapy (ACT); Hong Kong; Focused Acceptance Commitment Therapy (FACT); Psychological flexibility; Feasibility; Acceptability; Waitlist control group; Mental well-being
MeSH Terms: conditions — Neurodevelopmental Disorders; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Learning Disabilities; Chronic Disease; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Assigned by the investigator but not randomized
Who Masked: Outcomes Assessor
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACT Group (Experimental): 4-6 FACT consultation sessions, one weekly session, 45-60 mins per session. These sessions will be using online video conferencing platforms.
  Interventions: Behavioral: Focused Acceptance and Commitment Therapy
- Waitlist Control Group (Other): The waitlist control group participants will commence their intervention trial immediately after they complete their follow-up assessment.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: Focused Acceptance and Commitment Therapy — FACT aims to increase one's psychological flexibility so that one will not generate feelings of distress and suffering when confronted with painful life situations. The intervention of this study will follow the FACT principles laid out by Strosahl, Robinson and Gustavsson to increase parents' psychological flexibility. Three core processes influence one's psychological flexibility: awareness, openness, and engagement.
  The key objectives of each core process are:
  1. Awareness: Able to experience the present moment, able to take perspective on self
  2. Openness: Able to detach distressing private experiences and associated rules, able to take a non-judgemental, accepting stance towards painful material
  3. Engagement: Exhibits strong connection with values, able to sustain values-consistent action
  Arms: FACT Group
Other: Waitlist Control — The waitlist control group participants will commence their FACT intervention immediately after they complete their follow-up assessment.
  Arms: Waitlist Control Group

SUMMARY:
The purpose of the proposed non-randomized waitlist-controlled design study is to evaluate the feasibility, acceptability, and potential effectiveness of using a Videoconferencing-based Individual Focused Acceptance and Commitment Therapy (FACT) approach to enhance the mental well-being of parents of children with special healthcare needs (SHCN) over a three-month period after the intervention has taken place.

DETAILED DESCRIPTION:
Parents of children with special health care needs (SHCN) have always been under tremendous pressure to care for their children. The parental well-being, as well as family functioning, are at risk. In literature, there has been increasing evidence supporting the efficacy of Acceptance and Commitment Therapy (ACT) on mental health in different populations, including healthy individuals, parents, children and those with mental health problems. The previous studies done by the PI in using ACT for improving parental well-being and management have proven the intervention effective for Hong Kong parents. Her work showed that ACT training effectively enhanced the parental well-being of parents of children with asthma and autism spectrum disorder.

Though the result was promising, the previous clinical trials in Hong Kong showed a limited effect size. This is due to the need for extensive manpower in ACT intervention, yet there are very limited trained ACT interventionists in Hong Kong. On top of that, past interventions have failed to target impaired psychopathological processes as well as identify and determine which psychopathological processes require intervention in the first place. This study aims to overcome the limitations mentioned above. The proposed study will follow the model and principles of Focused Acceptance Commitment Therapy (FACT) to increase the psychological flexibility of parents of children with SHCN. FACT is a new model of brief therapy that is a highly condensed version of Acceptance and Commitment Therapy, which has been proven to be effective in the long term in improving one's mental well-being through increasing one's psychological flexibility. The time-limited and brief FACT intervention targets the impaired psychopathological processes and determines what process(es) need to work on first, which also eases the demand for ACT interventionists.

This study aims to evaluate the feasibility, acceptability, and possible effectiveness of Videoconferencing-based Individual Focused Acceptance and Commitment Therapy (FACT) in enhancing the mental health of parents of children with special healthcare needs (SHCN) by comparing the results to those of a waitlist control group. The study will assess the well-being of the participating parents before the intervention, immediately after the intervention and again three months later to determine the impact of the FACT intervention on their mental well-being.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese-speaking Hong Kong residents aged ≥21 years;
* living together with the child who is at preschool/school-age (3-9 years old);
* adopt the responsibility of taking care of the child;
* access to reliable Internet access via either computers and/or smartphones and be committed to maintaining internet access for the duration of the intervention

In addition, potential eligible parents who respond "yes" to any of the five validated screening questions in the Children with Special Health Care Needs (SHCN) Screener will then be asked the associated follow-up questions to determine whether the child possesses physical, neurodevelopmental/emotional problem(s) that has lasted for at least 12 months. Only children with a positive response(s) to ≥ 1 item in each of the associated follow-up questions will be classified as children with SHCN

Exclusion Criteria:

* Parents with cognitive deficiency, severe mental illness and/or disability conditions that interfere with their ability to comprehend the programme's content
* had substance/alcohol dependency problems,
* are pregnant;
* are less than six months postpartum

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Parental depressive symptoms | Change from baseline assessment to immediate and 3 months post-intervention
  The Patient Health Questionnaire (PHQ-9, 9-item, 4-point Likert scale) will be used to assess the frequency of the parents experiencing depressive symptoms in the past two weeks. The Chinese version of the PHQ-9 has demonstrated good internal consistency reliability (Cronbach's alpha = 0.86) and test-retest correlation coefficient.
Parental anxiety symptoms | Change from baseline assessment to immediate and 3 months post-intervention
  The Generalized Anxiety Disorder-7 (GAD-7, 7-item, 4-point Likert scale) will be used to measure the severity of anxiety symptoms. The Chinese version of the GAD-7 demonstrated good reliability and validity with a Cronbach's coefficient of 0.91.
Parental Stress | Change from baseline assessment to immediate and 3 months post-intervention
  The Parental Stress Scale (PSS, 18-item, 5-point scale) will assess parenting stress. A higher score represents a higher level of parental stress. The Chinese version of the PSS has demonstrated acceptable psychometric properties and is therefore suitable for use by researchers to assess the parental stress levels of Chinese parents.

SECONDARY OUTCOMES:
Parental Psychological Flexibility | Change from baseline assessment to immediate and 3 months post-intervention
  The PsyFlex (5-point Likert scale, 6 items) will be used to assess the six therapeutic processes in ACT, namely contacting the present moment, defusion, acceptance, self-as-context, values and committed action.

CONTACTS AND LOCATIONS:
Locations (5):
- Hong Kong (5):
  - Hong Kong Christian Service, Hong Kong
  - Hong Kong Federation of Youth Groups, Hong Kong
  - Hong Kong Young Women's Christian Association, Hong Kong
  - Yang Memorial Methodist Social Service, Hong Kong
  - Chinese University of Hong Kong, Shatin